CLINICAL TRIAL: NCT00581230
Title: An Evaluation Of The Rapid Airway Management Positioner (RAMP) In Obese Patients Undergoing Gastric Bypass Or Laparoscopic Gastric Banding (Lap-Band) Surgery
Brief Title: Evaluation of the Rapid Airway Management Positioner
Acronym: RAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chair - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-07-0067
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Endotracheal Intubation; Rapid Airway Management Positioner
Keywords: Endotracheal Intubation; Rapid Airway Management Positioner
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngoscopy without RAMP (Experimental): First, laryngoscopy will be preformed utilizing a traditional Macintosh size 4 blade laryngoscope. The view of the laryngeal aperture will be recorded, and a photo will be taken by the Airway Cam™.
  Interventions: Device: Laryngoscopy without RAMP
- Laryngoscopy with RAMP (Experimental): Next, the Rapid Airway Management Positioner (RAMP) will be positioned and inflated underneath the patient so that the patient is placed in the optimal sniffing position. The investigator will again perform laryngoscopy utilizing the same technique and the laryngeal view will be recorded.
  Interventions: Device: Laryngoscopy with RAMP

INTERVENTIONS:
Device: Laryngoscopy with RAMP — inflatable positioning ramp
  Arms: Laryngoscopy with RAMP
Device: Laryngoscopy without RAMP — Laryngoscopy without RAMP
  Arms: Laryngoscopy without RAMP

SUMMARY:
The purpose of this study is to determine if the Rapid Airway Management Positioner (RAMP, AirPal, Center Valley, PA) is a useful positioning device for direct laryngoscopy and tracheal intubation in obese patients undergoing gastric bypass or laparoscopic gastric banding surgery.

DETAILED DESCRIPTION:
The cannot intubate, cannot ventilate case is the most dangerous of situations, and being able to foresee, prevent, and prepare for such difficulties is the task of every anesthesiologist. Difficult mask ventilation is predicted by a number of factors, including obesity.1 Appropriate bag-and-mask ventilation necessitates a patent airway. An increased BMI is associated with a reduced posterior airway space behind the tongue's base as well as a quick development of hypoxemia from reduced functional residual capacity in improper mask ventilation.1 Proper head and neck positioning to establish the patent airway then is especially important.

There is an increased risk of difficult laryngoscopy among obese patients compared with subjects with normal body mass index.2,3 Optimal laryngeal view during laryngoscopy can be facilitated with proper head and neck positioning, including slight elevation of the head, neck flexion relative to the chest, and extreme atlanto-occipital extension.4 The "ramped" position, where the patient's ear is horizontally aligned with their sternal notch, has been found to be superior to the standard "sniffing" position, 7-cm occiput elevation, during direct laryngoscopy in morbidly obese patients.4

Additionally, there are increased difficulties and risks for tracheal intubation in obese patients versus normal-weight patients. Studies have found that chances for a successful first attempt at oral intubation decrease as patient weight increases.6,7 Improving visualization of laryngeal structures will increase the likelihood of successful tracheal intubation, as increasing the percentage of glottic opening is correlated with the number of intubation attempts, as well as the need for rescue intubation devices.8

It is estimated that endotracheal intubation is performed on approximately 8 million patients per year in the United States. Of these endotracheal intubations, approximately 80% are performed by direct laryngoscopy with transoral placement of the endotracheal tube (ET) into the trachea. There is fairly uniform reporting of the incidence of failed intubation in the literature; it occurs in approximately 0.05% or 1:2230 of surgical patients and in approximately 0.13% to 0.35%, or 1:750 to 1:280, of the obstetric patients.9,10 The incidence of unsuspected difficult intubation is estimated to be higher at 3%. One factor that contributes to difficult intubation is poor visualization, and difficult laryngoscopy is highly correlated with poor laryngeal exposure.11

The Rapid Airway Management Positioner (RAMP) is designed to optimize visualization during direct laryngoscopy by placing the patient into the proper head-elevated laryngoscopy position (HELP). In morbidly obese patients, achieving this position is important,12 and requires a great deal of support under the head and shoulders that could not be performed singlehandedly.13 The RAMP is an easy-to-use, quick device, taking an average of 56 seconds to place and inflate.14

The RAMP has great potential in obese patients. Pre-positioning also helps increase the desaturation safety period for morbidly obese patients.15 Rescue ventilation techniques are facilitated by the HELP position, when the head and neck are elevated above the chest and abdomen. The airway is therefore more isolated and easier to work with, and less positive airway pressure is needed when the weight of the abdomen is away from the diaphragm. Currently, placing a patient on top of stacked blankets is common and can create the HELP, or "ramped" position, 5 but also causes variable and unstable results. We suspect that by providing a better laryngeal view, the RAMP may help decrease the incidence of tissue trauma associated with intubation, and intubation may be achieved more quickly in a population that is known to be difficult.

ELIGIBILITY:
Inclusion Criteria:

* The 50 subjects will be adult surgical candidates age 18-80, ASA I-III, BMI > 30 kg/m2 presenting for gastric bypass or laparoscopic gastric banding surgery who require general anesthesia.

Exclusion Criteria:

* Patients will be excluded if it is determined that an awake intubation should be performed. Mallampati IV and ASA IV-V patients will also be excluded, as well as patients with unstable cervical, thoracic and/or lumbar fracture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A. Hagberg,, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients who presented to surgery and met inclusion criteria were enrolled in the study
Groups:
- Entire Study: All the patients first underwent mask ventilation and laryngoscopy with Macintosh size 4 blade laryngoscope without RAMP. Second, all patients underwent laryngoscopy with RAMP--the RAMP pillow was inflated for all patients and the ease of Mask ventilation and Cormack Lehane laryngoscopy view with Macintosh size 4 laryngoscope was recorded.
Period: Overall Study
Arm/Group | Entire Study
Started | 51
Laryngoscopy Without RAMP | 51
Laryngoscopy With RAMP | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Laryngoscopy Without RAMP, Then Laryngoscopy With RAMP: First, laryngoscopy was preformed utilizing a traditional Macintosh size 4 blade laryngoscope (without the Rapid Airway Management Positioner (RAMP)). The view of the laryngeal aperture was recorded, and a photo was taken by the Airway Cam™. Second, the Rapid Airway Management Positioner (RAMP) was positioned and inflated underneath the patient so that the patient was placed in the optimal sniffing position. The investigator again performed laryngoscopy utilizing the same technique, the second time with RAMP, and the laryngeal view was recorded.
Arm/Group | Laryngoscopy Without RAMP, Then Laryngoscopy With RAMP
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.76 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Ease of Mask Ventilation as Assessed by Han Class
Description: Grading Scale for Mask Ventilation as described by Han et al. (Anesthesiology. 2004 Jul;101(1):267) Grade 0. Ventilation by mask not attempted Grade 1. Ventilated by mask Grade 2. Ventilated by mask with oral airway/adjuvant with or without muscle relaxant Grade 3. Difficult ventilation (inadequate, unstable, or requiring two providers) with or without muscle relaxant Grade 4. Unable to mask ventilate with or without muscle relaxant
Time Frame: Time before intubation
Measure: Number; unit: participants
Groups:
- Laryngoscopy Without RAMP: In all participants, laryngoscopy was first performed utilizing a traditional Macintosh size 4 blade laryngoscope (without the Rapid Airway Management Postitioner (RAMP)). The view of the laryngeal aperture was recorded, and a photo was taken by the Airway Cam™.
- Laryngoscopy With RAMP: In this crossover study, all participants then received laryngoscopy with the Rapid Airway Management Positioner (RAMP) (immediately after Laryngoscopy without RAMP). The RAMP was positioned and inflated underneath the patient so that the patient was placed in the optimal sniffing position. The investigator again performed laryngoscopy utilizing the same technique, except that RAMP was used, and the laryngeal view was recorded.
Arm/Group | Laryngoscopy Without RAMP | Laryngoscopy With RAMP
Number analyzed (Participants) | 46 | 46
participants
  Grade 1 | 15 | 24
  Grade 2 | 18 | 15
  Grade 3 | 13 | 7
  Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: Laryngoscopy Without RAMP vs Laryngoscopy With RAMP; Test type: Superiority or Other; p = 0.0003, Wilcoxon signed rank test

2. Primary Outcome: Glottic View as Assessed by the Cormack and Lehane Classification
Description: Glottic view as described by Cormack and Lehane (Samsoon GL, Young JR. Difficult tracheal intubation: A retrospective study. Anesthesia 1987; 42:487), scored as follows- Grade 1. Full view of glottis Grade 2a. Partial view of glottis Grade 2b. Arytenoids or posterior portion of cords just visible Grade 3. Only the epiglottis visible Grade 4. Neither epiglottis nor glottis visible
Time Frame: before intubation
Measure: Number; unit: participants
Groups:
- Laryngoscopy Without RAMP: The Cormack Lehane grade view obtained with laryngoscopy when there was no RAMP pillow. In all participants, laryngoscopy was first performed utilizing a traditional Macintosh size 4 blade laryngoscope (without the Rapid Airway Management Postitioner (RAMP)). The view of the laryngeal aperture was recorded, and a photo was taken by the Airway Cam™.
- Laryngoscopy With RAMP: The Cormack Lehane grade glottic view obtained during laryngoscopy with inflated RAMP pillow. In all participants, laryngoscopy with the Rapid Airway Management Positioner (RAMP) was performed second (after Laryngoscopy without RAMP). The RAMP was positioned and inflated underneath the patient so that the patient was placed in the optimal sniffing position. The investigator again performed laryngoscopy utilizing the same technique, except that RAMP was used, and the laryngeal view was recorded.
Arm/Group | Laryngoscopy Without RAMP | Laryngoscopy With RAMP
Number analyzed (Participants) | 50 | 50
participants
  Grade 1 | 17 | 28
  Grade 2a | 11 | 13
  Grade 2b | 12 | 6
  Grade 3 | 7 | 2
  Grade 4 | 3 | 1
Statistical Analysis 1: Comparison: Laryngoscopy Without RAMP vs Laryngoscopy With RAMP; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test

ADVERSE EVENTS:
Groups:
- Entire Study: This is a crossover study, all the patients 1st underwent mask ventilation and laryngoscopy with Macintosh size 4 blade laryngoscope. After this, the RAMP pillow was inflated for all patients and the ease of Mask ventilation and Cormack Lehane laryngoscopy view with Macintosh size 4 laryngoscope was recorded.
Arm/Group | Entire Study
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

LIMITATIONS AND CAVEATS:
major limitations of the study was the lack of a blinded observer for the purpose of rating the laryngoscopic view & how easily, quickly & consistently this position can be achieved as well as to return the patient to a neutral position for surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No